CLINICAL TRIAL: NCT01729715
Title: Helping Young Children Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Splaingard, Prof. and Dir. of pediatric sleep medicine, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB12-00439
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Insomnia
Keywords: Pediatric; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Patient Portals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Internet (Experimental): Internet site that offers parents tips on promoting sleep in infants and toddlers
  Interventions: Behavioral: Internet
- DVD (Experimental): DVD that offers parents tips on promoting sleep in infants and toddlers
  Interventions: Behavioral: DVD
- No treatment (No Intervention)

INTERVENTIONS:
Behavioral: Internet
  Arms: Internet
Behavioral: DVD
  Arms: DVD

SUMMARY:
The investigators are conducting a randomized trial of behavioral treatments for young children with insomnia. The investigators are comparing the improvement in sleep patterns after families are given access to Internet sleep instructions compared to DVD sleep instructions.

ELIGIBILITY:
Inclusion Criteria:

* 6-36 months
* difficulties falling asleep or staying asleep
* DVD and internet access

Exclusion Criteria:

* Under 14 pounds
* Requires nighttime feeding or parental intervention for health reasons
* Chronic medical or psychological conditions such as asthma or autism
* Parents prefer co-sleeping

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Brief infant sleep questionnaire | 3 weeks
  infant sleep patterns and sleep problems

SECONDARY OUTCOMES:
Profile of mood states | 1 week
  parental mood in the past week
Pittsburgh sleep quality index | 1 month
  parental sleep patterns within the past month

CONTACTS AND LOCATIONS:
Overall Officials: Mark Splaingard, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States